CLINICAL TRIAL: NCT06942702
Title: Assesment of Postoperative Analgesic Efficacy of Preoperatively Applied Genicular Block on Total Knee Arthroplasty: A Randomized Controlled Study
Brief Title: Efficacy of Genicular Block on Total Knee Arthroplasty Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Mustafa Azizoğlu, Associated Professor, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MersinUgenicular
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Total Knee Anthroplasty; Genicular Nerves Block
Keywords: total knee arthroplasty; genicular block; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Passive Cutaneous Anaphylaxis; Acetaminophen; Diclofenac

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Genicular block group (Active Comparator): this group consists of the patients receiving genicular block preoperatively and they will be given morfin with PCA (Patient controlled analgesia) and paracetamol 3x1000 mg intravenous and diclofenac 75 mg intramuscular (if needed)
  Interventions: Drug: Genicular blocks (bupivakain); Drug: Patient Control Analgesia (PCA) Morphine group; Drug: Paracetamol (acetaminophen) + Diclofenac Sodium
- patients only given PCA-morfin postoperatively (Active Comparator): this group consists of the patients given morfin with PCA, paracetamol 3x1000 mg and diclofenac (if needed)
  Interventions: Drug: Patient Control Analgesia (PCA) Morphine group; Drug: Paracetamol (acetaminophen) + Diclofenac Sodium

INTERVENTIONS:
Drug: Genicular blocks (bupivakain) — Genicular block is a regional analgesic technique performed with USG
  Arms: Genicular block group
Drug: Patient Control Analgesia (PCA) Morphine group — this group consists of the patients no any intervention preoperatively and they will be given morfin with PCA (Patient controlled analgesia) and paracetamol 3x1000 mg intravenous and diclofenac 75 mg intramuscular (if needed)
  Other Names: PCA-M
Drug: Paracetamol (acetaminophen) + Diclofenac Sodium — All patients are given paracetamol (3x1000 mg) and diclofenac (if needed)

SUMMARY:
The aim of this study is to investigate the postoperative pain relieving effect of preoperative genicular block in total knee arthroplasty surgery. The main questions it aims to answer are:

1. Do visual analog scale (VAS) scores decrease in patients who underwent geniculate block?
2. Does opioid consumption decrease in patients who underwent geniculate block?

Researchers will compare postoperative pain in patients who received genicular block with those who did not.One group of patients will be administered 0.25% bupivacaine with the geniculate block method. The other group will not undergo any intervention. Both groups will be administered intravenous morphine for postoperative analgesia.

DETAILED DESCRIPTION:
Patients scheduled for knee arthroplasty will be randomly assigned into two groups. One group will receive a genicular nerve block prior to surgery without the administration of general anesthesia, while the other group will not undergo any interventional procedure. The genicular nerve block will be administered in three quadrants around the knee, with each injection consisting of 5 mL of 0.25% Marcaine. All injections will be performed by investigator MA. Patient assessments will be conducted by investigator MO. Postoperative intravenous analgesia will be provided to both groups.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for unilateral and primary total knee arthroplasty
* Older than 18 years of age

Exclusion Criteria:

* Younger than 18 years
* Bilateral knee arthroplasty
* Revision case of knee arthroplasty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-10-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale Measure | 0-48 hours
  VAS scores are assessed at 0th, 24th and 48th hours post operatively VAS score consists of 0-10 in numbers, the bigger the number the worse the pain
opioid consumption | 0-48 hours
  Morphine consumption is assesed by PCA

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Azizoglu, Associated Professor, Principal Investigator — Mersin university Faculty of Medicine, Department of Anesthesiology and Reanimation

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will not be shared due to ethical considerations and institutional policies on patient confidentiality.

REFERENCES:
- [Background] Wang T, Leng YF, Zhang Y, Kang YQ, Xue X, Zhang Y. [Preventive effects of ischemic postconditioning and penehyclidine hydrochloride on gastric against ischemia-reperfusion injury in rats]. Zhonghua Yi Xue Za Zhi. 2011 Apr 26;91(16):1130-5. Chinese. PMID 21609599